CLINICAL TRIAL: NCT04849273
Title: A Phase 1/2 Study of TPX-0131, A Novel Oral ALK Tyrosine Kinase Inhibitor in Subjects With ALK+ Advanced or Metastatic NSCLC
Brief Title: A Study of TPX-0131, a Novel Oral ALK Tyrosine Kinase Inhibitor, in Patients With ALK+ Advanced or Metastatic NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adverse change in the risk/benefit.
Sponsor: Turning Point Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA226-1036; CA226-1036 (Other: BMS Protocol ID); TPX-0131-01 (Other: Turning Point Therapeutics Protocol ID)
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Non Small Cell Lung Cancer; Non-Small Cell Lung Cancer; NSCLC; Advanced Solid Tumor; Metastatic Solid Tumor; ALK Gene Mutation
Keywords: Non Small Cell Lung Cancer; Non-Small Cell Lung Cancer; NSCLC; Advanced Non-Small Cell Lung Cancer; Advanced/metastatic disease; Lung cancer; Metastatic solid tumor; Advanced solid tumor; ALK gene fusion; ALK inhibitor; TPX-0131; ALK TKI; ALK Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms | interventions — TPX-0131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TPX-0131 (Experimental): The Phase 1 part of the study will determine the safety, tolerability, PK, MTD, and RP2D of TPX-0131.
  Interventions: Drug: TPX-0131

INTERVENTIONS:
Drug: TPX-0131 — Oral TPX-0131 tablets

SUMMARY:
A phase 1, first-in-human, open-label study to evaluate the safety, tolerability, PK, and efficacy of the novel ALK inhibitor TPX-0131 in pretreated subjects with ALK+ advanced or metastatic non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Phase 1 Dose Escalation: To evaluate the overall safety profile, efficacy of TPX-0131 in pretreated subjects with ALK+ advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 (or as required by local regulation).
* Histological or cytological confirmation of advanced/metastatic ALK+ NSCLC.
* Pretreated with up to three prior lines of an ALK TKI treatment, including at least one prior line of a second or third-generation ALK TKI (alectinib, brigatinib, ensartinib, or lorlatinib) in Phase 1.
* ECOG performance status ≤ 1.
* Existence of measurable or evaluable disease (according to Response evaluation criteria in solid tumors [RECIST v1.1] criteria).
* Subjects with asymptomatic CNS metastases and/or asymptomatic leptomeningeal carcinomatosis are eligible.
* Adequate organ function.

Exclusion Criteria:

* Major surgery within four weeks of the start of TPX-0131 treatment.
* Clinically significant cardiovascular disease
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) > 470 msec obtained from three ECGs and any factors that increase the risk of QTc prolongation or arrhythmic events
  * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG
* Known clinically significant active infections not controlled with systemic treatment (bacterial, fungal, viral including HIV positivity).
* Gastrointestinal disease or other malabsorption syndromes that would impact drug absorption.
* Subjects being treated with or anticipating the need for treatment with strong CYP3A4 inhibitors or inducers.
* Subjects with current or anticipated need for drugs that are sensitive CYP2C9 substrates with narrow therapeutic indices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Incidence of first cycle dose-limiting toxicities (DLTs) of TPX-0131 | Within 28 days of the first TPX-0131 dose for each patient
  Evaluate the safety and tolerability of TPX-0131
Define the Recommended Phase 2 Dose | Approximately 24 months
  Determine the maximum tolerated dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of TPX-0131

SECONDARY OUTCOMES:
Adverse events (AEs) | Approximately 34 months
  Evaluate the overall safety profile of TPX-0131

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- United States (7):
  - Local Institution - 2104, Orange, California
  - Local Institution - 2105, Aurora, Colorado
  - Local Institution - 2106, Boston, Massachusetts
  - Local Institution - 2108, Boston, Massachusetts
  - Local Institution - 2103, Hackensack, New Jersey
  - Local Institution - 2107, Nashville, Tennessee
  - Local Institution - 2102, Fairfax, Virginia
- Australia (4):
  - Local Institution - 6102, Blacktown, New South Wales
  - Local Institution - 6103, Heidelberg, Victoria
  - Local Institution - 6104, Melbourne, Victoria
  - Local Institution - 6101, Nedlands, Western Australia
- South Korea (4):
  - Local Institution - 6303, Seoul, Seoul-teukbyeolsi
  - Local Institution - 6301, Seoul
  - Local Institution - 6302, Seoul
  - Local Institution - 6304, Seoul

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm